CLINICAL TRIAL: NCT02415556
Title: Memory Advancement by Intranasal Insulin in Type 2 Diabetes
Brief Title: Memory Aid by Intranasal Insulin in Diabetes (MemAID)
Acronym: MemAID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry); Medtronic (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Vera Novak, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015P000064; 1R01DK103902-01A1 (NIH)
Record Dates: First submitted 2015-03-23; First posted 2015-04-14 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Intranasal Insulin; Placebo; Memory; Gait; Non diabetic older controls
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: 289 signed ICF.
  244 were randomized (115 T2DM adults and 129 non-DM controls).
  79 T2DM adults and 90 non-DM controls completed intervention (as of 4/23/2020)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Type 2 Diabetes Mellitus - Insulin (Experimental): 40 IU of regular human insulin once daily over 24 weeks
  Interventions: Drug: Regular Human Insulin
- Type 2 Diabetes Mellitus - Placebo (Placebo Comparator): Intranasal sterile saline once daily over 24 weeks
  Interventions: Drug: Placebo
- Control - Insulin (Experimental): 40 IU of regular human insulin once daily over 24 weeks
  Interventions: Drug: Regular Human Insulin
- Control - Placebo (Placebo Comparator): Intranasal sterile saline once daily over 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regular Human Insulin — Regular human insulin 40 IU daily over 24 weeks
  Other Names: Novolin R Novonordisk
  Arms: Control - Insulin; Type 2 Diabetes Mellitus - Insulin
Drug: Placebo — Intranasal sterile saline 40 IU daily over 24 weeks
  Other Names: Sterile normal saline
  Arms: Control - Placebo; Type 2 Diabetes Mellitus - Placebo

SUMMARY:
The main purpose of this study is to find the long-term effects of daily administration of 40 IU of intranasal insulin (INI) as compared to placebo (sterile saline) on cognition and memory in people with type 2 diabetes mellitus (DM), and non-diabetic controls over 24 weeks with a follow-up period for 24 weeks. Four groups will be tested: DM group treated with INI; DM group treated with placebo; control group treated with INI and the control group treated with placebo. The INI or placebo will be delivered into the nose. The investigators are interested to see whether INI can improve memory and cognition and blood flow in the brain in the type 2 DM group as compared to placebo and to the non-diabetic group over a long-term period.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial determining the long-term effects of intranasal insulin (INI) on cognition and memory in type 2 diabetes (DM) and non-DM groups. The investigators hypothesize that: 1) INI-treated adults with DM have better memory and functioning of specific cognitive domains and faster walking during a dual task than those treated with placebo and the control group; 2) Glycemic and insulin resistance and genetic markers for Alzheimer's disease (Apolipoprotein E4 [ApoE4]) may serve as predictors of positive responses to INI therapy; 3) INI treatment neither adversely affects systemic glycemic levels or the cardiovascular system nor causes weight gain.

Aim 1: To determine whether INI-treated type 2 DM adults have a) better memory and functioning of specific cognitive domains and b) faster dual-task gait speed and better daily living functioning than the placebo-treated and non-DM groups. Four groups will be tested: 60 DM subjects treated with insulin; 60 DM subjects treated with placebo; 45 control subjects treated with INI and 45 control subjects treated with placebo. These 210 patients are expected to complete treatment and 168 are expected to complete study by the study completion anticipated date.

The investigators will conduct a randomized, double-blind, placebo-controlled study in 120 older adults with type 2 DM and 90 non-DM controls examining whether 40 IU INI once daily over a 24-week period improves:

* Specific domains of visuospatial attention and memory, verbal learning (primary outcomes);
* Gait speed during a dual task (which is an excellent predictor of overall health), daily living functionality, and depression as compared to the DM group receiving sterile saline and the non-DM groups. The non-DM groups will provide reference of INI effects in a clinical phenotype of cognitive decline and insulin resistance that occurs with normal aging.

Aim 2: To identify a phenotype and long-term trajectory predicting clinically relevant response to INI therapy based on glycemic control, insulin resistance, endothelial and genetic markers.

1. The investigators will determine a phenotype predicting a clinically relevant response to INI therapy and identify time-dependent trajectories of INI effects on cognition in the DM group vs. the placebo and the non-DM groups. Clinical predictors will be based on associations between cognitive function and/or gait and demographic, glycemic control, insulin resistance, endothelial and genetic (ApoE4) measures.
2. The investigators will evaluate the dose-escalating trajectory of cognition, gait speed, and functionality during the 24 weeks of therapy and 24 weeks post-treatment and their dependence on the above-mentioned factors, and determine the time point when maximum effect was reached. INI therapy response is defined as a clinically relevant improvement on cognitive tests or in gait speed (as a continuous variable) or as responders vs. non-responders as compared to placebo within DM and non-DM groups (as a categorical variable).
3. MRI substudy: The investigators will explore the long-term INI effects on regional perfusion, vasodilatation, and resting functional connectivity in 40 DM subjects pre- and post- INI/placebo administration at the beginning and at the end of intervention and their relationships to cognitive outcomes. Regional perfusion and vasodilatation will be measured by pseudo-continuous arterial spin labeling (PCASL) MRI at 3 Tesla, and resting-state functional connectivity will be quantified from low-frequency (0.01-0.08 Hz) fluctuations (LFF) of the whole-brain blood-oxygen-level dependent (BOLD) functional Magnetic Resonance Imaging (fMRI).

Aim 3: To determine the long-term safety of INI vs. placebo with regard to glycemic control (fasting glucose, hemoglobin A1c [HbA1c], hypoglycemic episodes), vital signs, and body mass.

1. The investigators will obtain measurements of fasting glucose, insulin, vital signs, and body mass at baseline, 2-months, 4-months, and 6-months follow-up and keep weekly logs monitoring glucose and adverse events.
2. Safety substudy: In the first 20 DM patients treated with subcutaneous insulin, the investigators will conduct continuous glucose monitoring (CGM) OR 5 finger sticks/day (effective after 9/25/2017) for 1 week during baseline and during the first week of INI or placebo treatment to evaluate the INI effects on glycemic control, hypoglycemic episodes, and body weight.

This study may pave the way to potential treatment and/or cure of DM- and age-related cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50-85 years old
* Able to walk for 6 minutes
* Diabetes type 2 (DM) group: diagnosis and treatment for type 2 DM with non-insulin oral or injectable agents
* Non-DM group with similar age range as the DM group, non-diabetic fasting plasma glucose (<126 mg/dL) and hemoglobin A1c (HbA1c) (<6.5%)
* Participants capable of providing informed consent

Exclusion Criteria:

* Type 2 DM treated with insulin (since 9/25/2017)
* Type 1 DM
* Intolerance to insulin
* History of severe hypoglycemia
* Participants who have >1 asymptomatic and/or symptomatic episode of hypoglycemia (glucose < 54 mg/dL) during finger stick or plasma glucose (cut off value since 6/11/2018)
* Acute medical condition that required either hospitalization or surgery within the past 6 months (e.g., severe hypoglycemia, malignancies, myocardial infarction,stroke)
* Liver or renal failure or transplant
* Dementia (Mini Mental State Examination [MMSE] scores ≤20)
* Current recreational drug or alcohol abuse
* Serious systemic disease that would interfere with conduction of clinical trial (mild forms of neurological conditions e.g. Parkinson's Disease, autonomic neuropathy etc. would be allowed)
* Magnetic Resonance Imaging (MRI) substudy in 40 DM patients only: claustrophobia and implants incompatible with 3-Tesla MRI
* Safety substudy in 20 IDDM patients only: Insulin-treated type 2 diabetics with a C-peptide of <0.8 ng/mLd and fasting blood glucose >150 mg/dL will be excluded even without history of hypoglycemia during finger stick measurements.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Novak, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center; Peter Novak, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vera Novak, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lioutas VA, Alfaro-Martinez F, Bedoya F, Chung CC, Pimentel DA, Novak V. Intranasal Insulin and Insulin-Like Growth Factor 1 as Neuroprotectants in Acute Ischemic Stroke. Transl Stroke Res. 2015 Aug;6(4):264-75. doi: 10.1007/s12975-015-0409-7. Epub 2015 Jun 5. PMID 26040423
- [Background] Lioutas VA, Novak V. Intranasal insulin neuroprotection in ischemic stroke. Neural Regen Res. 2016 Mar;11(3):400-1. doi: 10.4103/1673-5374.179040. No abstract available. PMID 27127468
- [Background] Zhang H, Hao Y, Manor B, Novak P, Milberg W, Zhang J, Fang J, Novak V. Intranasal insulin enhanced resting-state functional connectivity of hippocampal regions in type 2 diabetes. Diabetes. 2015 Mar;64(3):1025-34. doi: 10.2337/db14-1000. Epub 2014 Sep 23. PMID 25249577
- [Background] Galindo-Mendez B, Trevino JA, McGlinchey R, Fortier C, Lioutas V, Novak P, Mantzoros CS, Ngo L, Novak V. Memory advancement by intranasal insulin in type 2 diabetes (MemAID) randomized controlled clinical trial: Design, methods and rationale. Contemp Clin Trials. 2020 Feb;89:105934. doi: 10.1016/j.cct.2020.105934. Epub 2020 Jan 7. PMID 31923471
- [Background] Trevino JT, Quispe RC, Khan F, Novak V. Non-Invasive Strategies for Nose-to-Brain Drug Delivery. J Clin Trials. 2020;10(7):439. Epub 2020 Dec 10. PMID 33505777
- [Result] Novak V, Mantzoros CS, Novak P, McGlinchey R, Dai W, Lioutas V, Buss S, Fortier CB, Khan F, Aponte Becerra L, Ngo LH. MemAID: Memory advancement with intranasal insulin vs. placebo in type 2 diabetes and control participants: a randomized clinical trial. J Neurol. 2022 Sep;269(9):4817-4835. doi: 10.1007/s00415-022-11119-6. Epub 2022 Apr 28. PMID 35482079
- [Derived] Isaza-Pierrotti DF, Khan F, Novak P, Lioutas V, Mantzoros CS, Ngo LH, Novak V. Dropout risk and effectiveness of retention strategies in the Memory Advancement by Intranasal Insulin in Type 2 Diabetes (MemAID) Clinical Trial. Contemp Clin Trials. 2023 Feb;125:107057. doi: 10.1016/j.cct.2022.107057. Epub 2022 Dec 17. PMID 36539060
- [Derived] Trevino JA, Novak P. TS-HDS and FGFR3 antibodies in small fiber neuropathy and Dysautonomia. Muscle Nerve. 2021 Jul;64(1):70-76. doi: 10.1002/mus.27245. Epub 2021 Apr 15. PMID 33792960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two hospital sites. The study was activated by IRB on 4/1/42015. The first participant was enrolled (signed ICF) at BIDMC on 10/6/2015 and at BWH 6/22/2017 and the last participant was enrolled in December 2019.
Pre-assignment Details: Of 668 screened participants, 289 signed ICF( enrolled), 244 were randomized to INI or placebo treatment, 223 completed baseline and were analyzed.
Period: Overall Study
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Started | 57 | 58 | 65 | 64
Completed | 32 | 37 | 43 | 44
Not Completed | 25 | 21 | 22 | 20
Not completed — Adverse Event | 3 | 4 | 2 | 4
Not completed — Lost to Follow-up | 4 | 5 | 4 | 1
Not completed — Withdrawal by Subject | 13 | 4 | 14 | 12
Not completed — Physician Decision | 1 | 3 | 1 | 2
Not completed — Censored - study completion | 4 | 5 | 1 | 0
Not completed — Family-related issues | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of 244 randomized participants, 223 participants completed baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo | Total
Number analyzed (Participants) | 51 | 55 | 58 | 59 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.5) | 65.7 (8.7) | 66.1 (9.2) | 66.1 (9.2) | 65.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 29 | 31 | 109
  Male | 27 | 30 | 29 | 28 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 1 | 3 | 13
  Not Hispanic or Latino | 48 | 49 | 57 | 56 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 16 | 4 | 6 | 34
  White | 36 | 34 | 52 | 51 | 173
  More than one race | 3 | 4 | 0 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 55 | 58 | 59 | 223

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed Normal Walk (cm/s).
Description: Gait speed normal walk (cm/s) - difference between Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo, Control - Insulin vs. Control - Placebo.
Time Frame: Measured at baseline, on-treatment (V2-intervention week 1, V4 week 8, V6 week 16, V8 week 24) and post-treatment (V9-week 25, V10-week 32, V11-week 40, V12-week 48).
Population: Intention-to-treat analyses (Model 1) included data from 223 randomized subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 51 | 55 | 58 | 59
cm/s
  Baseline | 112.23 (22.94) | 103.42 (21.04) | 121.58 (21.87) | 119.51 (15.61)
  On-treatment average | 112.43 (22.03) | 105.83 (21.27) | 123.89 (23.36) | 119.44 (18.60)
  Post-treatment average | 113.12 (19.60) | 107.27 (23.16) | 124.79 (24.75) | 120.50 (19.33)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; We set type-I error rate at 0.05, power of 0.80 or above, effect size of 15% improvement due to INI, and obtained n=120 for the DM group (60 DM-INI; 60 DM-Placebo) and n=90 for the Control group (45 Control-INI; 45 Control-Placebo) yielding 210 patients with data at the end of the treatment period; Test type: Other — A spatial power variance-covariance structure was used to model within-subject correlated measurements where the number of days from the baseline visit was used as the power of the autoregressive correlation coefficient. Each efficacy and safety outcome variable was modeled separately. The independent variables included: 4 treatment groups, TIMEG (baseline, on-treatment and post-treatment period), TIMEG * treatment group.; an average number of treatment days; subjects as random effects; p = 0.025, Mixed Models Analysis — Mixed model p-value represents on-treatment difference between between Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo; Mean Difference (Final Values) = 6.52, 95% CI 2-sided [0.81 to 12.23]
Statistical Analysis 2: Comparison: Control - Insulin vs Control - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The independent variables in the model included a four-level indicator variable for the four treatment groups, a three-level time indicator variable (TIMEG) representing baseline, on-treatment and post-treatment period and an interaction term between TIMEG and treatment group. An average number of treatment days at each assessment visit was used as a continuous repeated variable and subjects were included as random effects. Each efficacy and safety outcome variable was modeled separately; p = 0.051, Mixed Models Analysis — Mixed model p-value represents on-treatment difference between between Control - Insulin vs. Control - Placebo; Mean Difference (Final Values) = 5.28, 95% CI 2-sided [-0.03 to 10.60]

2. Primary Outcome: Gait Speed Dual-task (cm/s).
Description: Gait speed dual-task (cm/s) - walking and counting backwards (subtracting 7) difference between Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo, Control - Insulin vs. Control - Placebo.
Time Frame: as for outcome 1
Population: Intention-to-treat analyses (Model 1) included data from 223 randomized subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 51 | 55 | 58 | 59
cm/s
  Baseline | 104.23 (23.30) | 93.18 (22.71) | 109.44 (24.40) | 110.24 (16.50)
  On-treatment average | 105.34 (23.59) | 98.27 (22.39) | 114.66 (25.11) | 112.58 (17.99)
  Post-treatment average | 108.77 (20.49) | 102.22 (21.02) | 117.29 (26.73) | 113.08 (20.60)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.31, 95% CI 2-sided [2.33 to 14.29]
Statistical Analysis 2: Comparison: Control - Insulin vs Control - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.342, Mixed Models Analysis — Mixed model p-value represents on-treatment difference between between Control - Insulin vs. Control - Placebo; Mean Difference (Final Values) = 2.71, 95% CI 2-sided [-2.90 to 8.32]

3. Primary Outcome: Executive Function Composite z Score
Description: The executive function composite score was calculated as a sum of Paired Associates Learning (PAL) and Spatial Working Memory (SWM) z-scores (range -2 to +2, 0 indicates the mean; higher score indicates worse outcome). Paired Associates Learning - raw score of Total Errors Adjusted (range 0-120) was converted to z-score. Spatial Working Memory - raw score SWM-Between Errors (range 0-42) and raw score of SWM-Strategy (range 8-56) were converted to z-scores. Executive function composite scores were compared between:
  Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo, Control - Insulin vs. Control - Placebo.
Time Frame: as for outcome 1
Population: Intention-to-treat analyses (Model 1) included data from 223 randomized subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 51 | 55 | 58 | 59
units on a scale
  Baseline | 0.84 (2.08) | 1.40 (2.30) | 0.46 (2.25) | 0.66 (2.22)
  On-treatment average | 0.13 (2.11) | 0.47 (2.48) | -0.51 (2.56) | 0.14 (2.34)
  Post-treatment average | -0.19 (2.16) | -0.11 (2.44) | -1.08 (2.38) | -0.31 (2.43)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.144, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.87 to 0.13]
Statistical Analysis 2: Comparison: Control - Insulin vs Control - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.008, Mixed Models Analysis — Mixed model p-value represents on-treatment difference between between Control - Insulin vs. Control - Placebo; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.11 to -0.16]

4. Primary Outcome: Verbal Memory Composite z Score
Description: Verbal memory composite score was calculated as the sum of Verbal Recognition Memory (VRM) z scores ( 0 indicates the mean; lower score indicates worse outcome). VRM- Free Recall raw score (range 0-12), immediate and delayed VRM-Recognition raw score (range 0-24) were converted to z-scores. Verbal memory composite scores were compared between Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo, Control - Insulin vs. Control - Placebo.
Time Frame: as for outcome 1
Population: Intention-to-treat analyses (Model 1) included data from 223 randomized subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 51 | 55 | 58 | 59
score on a scale
  Baseline | -0.74 (2.72) | -0.89 (3.02) | 0.07 (2.69) | -0.22 (2.33)
  On-treatment average | -0.16 (2.31) | -0.50 (2.20) | 0.34 (2.16) | -0.01 (2.34)
  Post-treatment average | 0.05 (2.21) | -0.24 (1.98) | 1.01 (1.82) | 0.23 (2.56)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.149, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.13 to 0.83]
Statistical Analysis 2: Comparison: Control - Insulin vs Control - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.134, Mixed Models Analysis — Mixed model p-value represents on-treatment difference between between Control - Insulin vs. Control - Placebo; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.11 to 0.80]

5. Secondary Outcome: Fasting Plasma Glucose (mg/dL).
Description: Long-term safety measure of fasting plasma glucose difference between Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo, Control - Insulin vs. Control - Placebo.
Time Frame: as for outcome 1
Population: Intention-to-treat analyses (Model 1) included data from 223 randomized subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 51 | 55 | 58 | 59
mg/dL
  Baseline | 138.63 (44.60) | 141.25 (51.15) | 92.07 (7.72) | 90.54 (7.71)
  On-treatment average | 140.47 (44.71) | 132.18 (39.45) | 90.11 (7.97) | 89.61 (9.33)
  Post-treatment average | 143.28 (51.69) | 140.34 (42.49) | 90.05 (7.62) | 91.94 (12.56)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = 10.29, 95% CI 2-sided [1.00 to 19.58]
Statistical Analysis 2: Comparison: Control - Insulin vs Control - Placebo; See primary aims; Test type: Other — See primary aims; p = 0.607, Mixed Models Analysis — See primary aims; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [-6.22 to 10.63]

6. Secondary Outcome: Weight (kg).
Description: Long-term safety measure of weight difference between Type 2 Diabetes Mellitus - Insulin vs. Type 2 Diabetes Mellitus - Placebo, Control - Insulin vs. Control - Placebo.
Time Frame: as for outcome 1
Population: Intention-to-treat analyses (Model 1) included data from 223 randomized subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 51 | 55 | 58 | 59
kg
  Baseline | 90.36 (21.80) | 90.96 (20.03) | 75.89 (14.19) | 76.40 (17.76)
  On-treatment average | 88.44 (19.75) | 93.79 (18.50) | 75.97 (13.43) | 77.14 (18.34)
  Post-treatment average | 90.41 (19.82) | 92.59 (19.23) | 76.15 (13.58) | 78.18 (19.21)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; See primary aims; Test type: Other — See primary aims; p = 0.576, Mixed Models Analysis — See primary aims; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-9.50 to 5.29]
Statistical Analysis 2: Comparison: Control - Insulin vs Control - Placebo; See primary aims; Test type: Other — See primary aims; p = 0.802, Mixed Models Analysis — See primary aims; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-7.58 to 5.87]

7. Other Pre Specified Outcome: Cerebral Blood Flow on Magnetic Resonance Imaging (MRI).
Description: Difference in regional cerebral blood flow in right medial prefrontal cortex (MPFC) was measured by pseudo-continuous arterial spin labeling (PCASL) MRI at 3 Tesla in 8 Type 2 Diabetes Mellitus - Insulin participants and 3 Type 2 Diabetes Mellitus - Placebo participants only.
Time Frame: At baseline and at V8 (week 24) the last intervention.
Population: MRI at 3 Tesla performed in 8 Type 2 Diabetes Mellitus - Insulin participants and 3 Type 2 Diabetes Mellitus - Placebo participants only.
Measure: Mean (Standard Deviation); unit: 50ml/100g/min
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
Number analyzed (Participants) | 8 | 3 | 0 | 0
50ml/100g/min
  Baseline | 86.40 (6.71) | 95.23 (0.52) |  |
  End of treatment | 92.68 (6.77) | 92.73 (0.98) |  |
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus - Insulin vs Type 2 Diabetes Mellitus - Placebo; Test type: Equivalence — CBF and vasoreactivity maps were analyzed on a voxel-by-voxel basis using Statistical non-Parametric Mapping (SnPM, http://www.sph.umich.edu/ni-stat/SnPM/), voxel-level threshold p < 0.005; p = 0.03, Voxel-Based Morphometry

ADVERSE EVENTS:
Time Frame: 48 weeks.
Arm/Group | Type 2 Diabetes Mellitus - Insulin | Type 2 Diabetes Mellitus - Placebo | Control - Insulin | Control - Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/55 | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/55 | 2/58 | 3/59
Other Adverse Events (participants affected / at risk) | 31/51 | 37/55 | 33/58 | 33/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 2 Diabetes Mellitus - Insulin (N=51) | Type 2 Diabetes Mellitus - Placebo (N=55) | Control - Insulin (N=58) | Control - Placebo (N=59)
Cardiac disorders - Others, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 2 Diabetes Mellitus - Insulin (N=51) | Type 2 Diabetes Mellitus - Placebo (N=55) | Control - Insulin (N=58) | Control - Placebo (N=59)
Flu-like symptoms (General disorders) | 13 (17) | 11 (12) | 8 (12) | 17 (17)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 3 (4) | 4 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (8) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 3 (4) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (5) | 3 (6) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02415556/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT02415556/ICF_000.pdf